CLINICAL TRIAL: NCT02201407
Title: Open, Multicenter, Local, Non-Randomized, Non-Interventional Study in Patients With Chronic Hepatitis B Receiving Therapy With PEGASYS® (Peginterferon Alfa-2a 40kD) - PRO B
Brief Title: An Observational Study in Participants With Chronic Hepatitis B (CHB) Receiving Therapy With Peginterferon Alfa-2a 40 Kilodaltons (kD) (PEGASYS) - The PRO B Study
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29062
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CHB Participants Treated With Peginterferon alfa-2a: As this is an observational study, treatment schedule will be at the clinician's discretion in accordance with local labeling and not directed by the protocol. Participants with CHB who are receiving peginterferon alfa-2a treatment according to standard of care, current summary of product characteristics, and in line with the local labeling will be followed for the duration of treatment with peginterferon alfa-2a (48 weeks) and up to 24 weeks after peginterferon alfa-2a treatment (72 weeks in total).
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a treatment according to standard of care, current summary of product characteristics and in line with the local labeling.
  Other Names: PEGASYS

SUMMARY:
This open--label, multicenter, national observational study will investigate the effectiveness of standard of care treatment with peginterferon alfa-2a in participants with chronic hepatitis B (CHB). Participants who have never received any hepatitis B virus (HBV) treatment and participants previously treated with nucleos(t)ide analogs (NAs) are qualified for enrollment. The observation period is 48 weeks (peginterferon alfa--2a standard of care treatment) and for up to 24 weeks thereafter (72 weeks in total).

ELIGIBILITY:
Inclusion Criteria:

* HBeAg positive or HBeAg negative serologically proven CHB with or without cirrhosis (histologically verified at some point in the past)
* Baseline HBV DNA greater than (>) 2000 IU/mL
* Elevated serum ALT > upper limit of normal (ULN)
* Participants treated with previous NAs therapy are eligible for this study

Exclusion Criteria:

* Participants who have contraindications for peginterferon alfa-2a in accordance with the approved summary of product characteristics (for example, severe psychiatric diseases, immunological diseases, severe hepatic dysfunction or decompensated cirrhosis of the liver severe retinopathy or thyroid dysfunction, autoimmune hepatitis, history of severe pre-existing cardiac disease, or hypersensitivity to the active substance, to alpha interferons, or to any of the excipients)
* Participants with ALT > 10 times of ULN or evidence of hepatocellular carcinoma
* Participants with serological evidence of co-infection with hepatitis A virus, hepatitis C virus, human immunodeficiency virus, or hepatitis D virus
* Participants with decompensated liver disease
* Pregnant or breast-feeding women
* A history of liver transplantation or planned for liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants receiving treatment for CHB with peginterferon alfa-2a according to standard of care and in line with the current summary of product characteristics and local labeling who have no contraindication to peginterferon alfa-2a therapy as per the local label. Target population are naïve participants (who have never received any HBV treatment) and previously treated participants with NAs.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Hepatitis B Envelope Antigen (HBeAg)- Positive CHB Achieving Sustained Immune Control | Week 72
  Sustained immune control is defined as a combined response: post-treatment HBeAg seroconversion, and HBV deoxyribonucleic acid (DNA) levels less than (<) 2000 international units per milliliter (IU/mL), and alanine aminotransferase (ALT) normalization.
Percentage of Participants With HBeAg-Negative CHB Achieving Sustained Immune Control | Week 72
  Sustained immune control is defined as a combined response: HBV DNA levels <2000 IU/mL and ALT normalization.

SECONDARY OUTCOMES:
Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Seroclearance or Seroconversion | Week 72
Percentage of Participants With HBeAg-Positive CHB Achieving Combined Response | Week 48
  Combined response is defined as: post-treatment HBeAg seroconversion, HBV DNA levels <2000 IU/mL, and ALT normalization.
Percentage of Participants With HBeAg-Negative CHB Achieving Combined Response | Week 48
  Combined response is defined as: HBV DNA levels <2000 IU/mL and ALT normalization.
Percentage of Participants With Serious Adverse Events (SAEs) and Non-SAEs | Up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Serbia (6):
  - Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Center of Serbia; Institute For Infectious Diseases, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinic for Infectious Diseases CC Kragujevac, Kragujevac
  - Clinic for Infectious Diseases CC Nis, Niš
  - Clinical Center Vojvodine; Clinic for Infectious Diseases; Clinic for Hematology, Novi Sad